CLINICAL TRIAL: NCT06650046
Title: Study on Topping-off Technique for Treating Lumbar Degenerative Diseases
Brief Title: Study on Topping-off Technique for Treating LDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Topping-off Technique
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Degenerative Disease
Keywords: Topping-off technique

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topping-off group (Experimental): Topping-off group Patients who have undergone the Topping-off surgery for lumbar spondylosis and have complete follow-up data and meet the standards completed at the First Affiliated Hospital of Shandong First Medical University.
  Interventions: Procedure: Topping-off Group; Procedure: Fusion Group
- Fusion group (Active Comparator): Patients who have undergone lumbar spine fusion surgery due to lumbar spondylosis and meet the standards and have complete follow-up data completed at the First Affiliated Hospital of Shandong First Medical University.
  Interventions: Procedure: Topping-off Group; Procedure: Fusion Group

INTERVENTIONS:
Procedure: Topping-off Group — Topping-off group Patients who have undergone the Topping-off system insertion surgery for lumbar spondylosis and have complete follow-up data and meet the standards completed at the First Affiliated Hospital of Shandong First Medical University.
  Fusion group Patients who have undergone lumbar spine fusion surgery due to lumbar spondylosis and meet the standards and have complete follow-up data completed at the First Affiliated Hospital of Shandong First Medical University.
Procedure: Fusion Group — Topping-off group Patients who have undergone the Topping-off system insertion surgery for lumbar spondylosis and have complete follow-up data and meet the standards completed at the First Affiliated Hospital of Shandong First Medical University.
  Fusion group Patients who have undergone lumbar spine fusion surgery due to lumbar spondylosis and meet the standards and have complete follow-up data completed at the First Affiliated Hospital of Shandong First Medical University.

SUMMARY:
Lumbar degenerative disease is a common disease among middle-aged and elderly people as well as those who sit for a long time, mainly manifested as symptoms such as lower back pain, stiffness, and numbness in the lower limbs. Traditional surgical treatments such as lumbar fusion can alleviate symptoms, but may lead to complications such as adjacent segment degeneration. Therefore, exploring safer and more effective treatment methods is of great significance. Topping off technique, as a new treatment method, combines the advantages of interbody fusion and dynamic fixation, aiming to reduce the pressure on the intervertebral disc at the surgical site, promote the repair of diseased intervertebral discs, while preserving partial mobility of the lumbar spine.The aim of this study is to evaluate the clinical efficacy and imaging changes of Topping off technique in the treatment of lumbar degenerative diseases. The Topping off technique combines posterior lumbar interbody fusion (PLIF) and Wallis interspinous dynamic fixation device implantation. Through prospective clinical trials, its therapeutic effect on patients with continuous double segment lumbar degenerative diseases was observed. The study included patients who underwent surgery for degenerative lumbar diseases in L4-5 and L5-S1, who were treated with two-stage fusion surgery and Topping off technique, respectively. Follow up was conducted before and after surgery, with an average follow-up time of 24 months. Evaluate preoperative and postoperative efficacy using Oswestry Disability Index (ODI), Pain Visual Analog Scale (VAS), and Japanese Orthopaedic Association (JOA) lumbar spine function score, and calculate recovery rate. At the same time, X-ray and MRI images were used to detect the overall range of motion (L2~S1ROM) of the lumbar spine, the range of motion (ROM) of the Wallis device inserted segments, the intervertebral disc height index (DHI), and the relative signal intensity of the nucleus pulposus (RSI) of the intervertebral disc.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical efficacy and imaging changes of Topping off technique in the treatment of lumbar degenerative diseases. The Topping off technique combines posterior lumbar interbody fusion (PLIF) and Wallis interspinous dynamic fixation device implantation. Through prospective clinical trials, its therapeutic effect on patients with continuous double segment lumbar degenerative diseases was observed. The study included patients who underwent surgery for degenerative lumbar diseases in L4-5 and L5-S1, who were treated with two-stage fusion surgery and Topping off technique, respectively. Follow up was conducted before and after surgery, with an average follow-up time of 24 months. Evaluate preoperative and postoperative efficacy using Oswestry Disability Index (ODI), Pain Visual Analog Scale (VAS), and Japanese Orthopaedic Association (JOA) lumbar spine function score, and calculate recovery rate. At the same time, X-ray and MRI images were used to detect the overall range of motion (L2~S1ROM) of the lumbar spine, the range of motion (ROM) of the Wallis device inserted segments, the intervertebral disc height index (DHI), and the relative signal intensity of the nucleus pulposus (RSI) of the intervertebral disc.

ELIGIBILITY:
Inclusion Criteria:

* The patient's clinical manifestations, physical examination, and imaging data all support the diagnosis of degenerative lumbar spondylosis.
* Those who have undergone strict and formal conservative treatment for at least 3 months before surgery and have no significant improvement in symptoms.
* Preoperative imaging examination showed L4-5 and L5-S1 responsible segment protrusion or protrusion leading to segment stenosis.
* Surgeries are performed by the same chief surgeon.

Exclusion Criteria:

* Lumbar instability, lumbar spondylolisthesis above grade II.
* Patients with severe osteoporosis, tuberculosis, or tumors.
* Systemic diseases that affect surgical treatment and medication, such as heart disease, liver disease, and kidney disease.
* Patients with mental illness, poor compliance, and inability to cooperate in completing follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS | 2 Years
  The visual analog scale (VAS) is used for pain assessment. It is widely used in clinical practice in China, and the basic method is to use a vernier ruler with a length of about 10cm, marked with 10 scales on one side, with both ends
  - Page 3 of 5 [DRAFT] - The visual analog scale (VAS) is used for pain assessment. It is widely used in clinical practice in China, and the basic method is to use a vernier ruler with a length of about 10cm, marked with 10 scales on one side, with both ends marked as "0" and "10" respectively. A score of 0 indicates painlessness, and a score of 10 represents the most severe pain that cannot be tolerated.
  pain that cannot be tolerated.
JOA | 2 Years
  The Japanese Orthopaedic Association Scores (JOA) is a neurological function scoring system recommended by the Japanese Orthopaedic Association, which includes four parts: upper limb motor function, lower limb motor function, sensory and bladder function, with a total score of 29 points. The lower the score, the more severe the neurological dysfunction.
Cobb angle of surgical space and adjacent space in neutral position, over extension and over flexion position | 2 Years
  Cobb angle of surgical space and adjacent space in neutral position, over extension and over flexion position

SECONDARY OUTCOMES:
Lumbar spine overall range of motion (L2~S1ROM) | 2 Years
  Lumbar spine overall range of motion (L2~S1ROM)
Wallis device insertion segment mobility (ROM) | 2 Years
  Wallis device insertion segment mobility (ROM)
Intervertebral Disc Height Index (DHI) | 2 Years
  Intervertebral Disc Height Index (DHI)

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Xuan Zhang, Ph.D/MD, Study Chair — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No